CLINICAL TRIAL: NCT06508203
Title: The Effect of Piroxicam Addition During Arthrocentesis on Mouth Opening and Postoperative Pain in the Management of Internal Derangement in Female Patients. (A Randomized Clinical Trial)
Brief Title: The Effect of Piroxicam Addition During Arthrocentesis on Mouth Opening and Postoperative Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 953mscfdasu
Record Dates: First submitted 2024-07-13; First posted 2024-07-18 (Actual); Last update posted 2024-07-18 (Actual); Status verified 2024-01

CONDITIONS: Temporomandibular Joint Disorders
MeSH Terms: conditions — Temporomandibular Joint Disorders | interventions — Arthrocentesis; Piroxicam

STUDY DESIGN:
Intervention Model Description: two arm randomized clinical trial with study group and positive control
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: triple masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): 20 patients will be treated by arthrocentesis with lactate ringer followed by injection with piroxicam 2 ml (40mg) (study group).
  Interventions: Procedure: arthrocentesis with lactate ringer followed by injection with piroxicam 2 ml (40mg)
- control (Active Comparator): 20 patients will be treated by arthrocentesis with lactate ringer only (control group).
  Interventions: Procedure: arthrocentesis with lactate ringer only

INTERVENTIONS:
Procedure: arthrocentesis with lactate ringer only — classical arthrocentesis with lactate ringer only (control group).
  Arms: control
Procedure: arthrocentesis with lactate ringer followed by injection with piroxicam 2 ml (40mg) — classical arthrocentesis with lactate ringer followed by injection with piroxicam 2 ml (40mg)
  Arms: study group

SUMMARY:
TMDs is an ancient condition discovered thousands of years ago. Historians state that the ancient Egyptians were the first who managed TMDs. They manually treated joint dislocation by away similar to ours nowadays. In the fifth century B.C, Hippocrates described technique for management of mandibular dislocation followed by concerns similar to fixation. At first the surgical management was performed to treat ankylosis and recurrent dislocation. The first surgical repositioning of articular disc done by Annandale in 1887. Lanz, Pringle and Wakeley were the first surgeons who did surgical removal of articular disc in the early 1900s. Their purpose was to manage signs and symptoms of TMDs which is pain, trismus clicking and limitation of movement. In addition, in the late 1800s, dentists' concerns changed toward occlusal adjustment during replacement of natural teeth and prosthetics procedures to avoid TMDs. At the beginning of the 20th century, dentists and otolaryngologists were ascribing head, face, ear, and jaw symptoms to pressure atrophy of the meniscus, glenoid fossa, and cranium as a result of the loss of posterior teeth. However, it was not until 1934 that "TMJ" became universally recognized when Costen, an otolaryngologist, published his discoveries claiming that pain in and around the jaw. Symptoms of Costen syndrome includes impaired hearing, ear pain, tinnitus, dizziness, burning sensation in throat and tongue, headache and trismus. Costen stated that the previous symptoms occur as a result of atrophic or perforated menisci, compression of Eustachian tube, erosion of bone of glenoid fossa and irritation of temporal and corda tympani nerve. On the other hand, in 1926, McCollum founded the Gnathological Society of California. Stallard had already coined the word "gnathology" in 1924. Gnathology is the harmonization of occlusal and inter jaw relationship for optimum dental and TMDs treatment. In addition, Kingsley in 1887 was the first to publish information on intraoral appliances (occlusal splint). Thompson in 1940s considered a leader in mandibular repositioning and rest position intraoral appliances. Shore advanced his concept of auto repositioning the mandible in the 1950s to fully seat the condyle, and Sears reintroduced pivot appliances in the late 1950s to "unload the condyle." Ramjford popularized the use of occlusal splints in the 1960s on the basis of his electromyographic. All the previous work depends on gnathonic concepts. Also, in 1960s Gelb introduced mandibular orthopedic repositioning appliance (MORA) to adjust condyle in its normal position. It has one risk which is irreversible changes in occlusal occurred with full time wear. By the late 1940s Schwartz explained the importance of masticatory musculature and specifically emotional tension as a primary etiologic factor for TMDs. Regional and referred pain of myofascial origin was considered to have a great effect on these conditions. It could be treated by physical medicine. By 1996 the AAOP published new guidelines on orofacial pain classification assessment and management. In addition, Guidelines for TMDs which are:

1. Temporomandibular disorders (TMD) are defined as a collective term consists of a number of clinical problems that include the muscles of mastication, the temporomandibular joint and surrounding structures, or both.
2. Temporomandibular disorders (TMD) are characterized by the following clinical presentation: pain in the muscles of mastication, the preauricular area and/or TMJ that is usually aggravated by manipulation or function; in addition to limited range of motion, abnormal mandibular movement, and locking of the joint. In addition to clicking
3. Common complaints as headache, earache, and orofacial pain, as well as masticatory muscle hypertrophy and abnormal occlusal wearing addition to tinnitus, ear fullness.
4. Cross-sectional epidemiologic studies of a specific nonpatient population show that approximately 75% have at least one sign and approximately 33% have at least one symptom; however, only 5% to 7% are estimated to need treatment. Prevalence data from clinical reports reveal a female to male ratio of 4:1 to 6:1 in persons seeking care, primarily in the second through the fourth decade of life.1 One of the recent treatment modalities of TMJ problems and TMDs is arthrocentesis (joint lavage).

DETAILED DESCRIPTION:
Materials and Methodology Design of the study: Randomized controlled Trial (RCT) Site of the study: department of oral and maxillofacial surgery faculty of dentistry Ain shams university Criteria of inclusion: study done on 40 patients have the following criteria

1. Age range 18-60 years both gender
2. Patient have gone on noninvasive therapy (occlusal stent) for three months without good prognosis
3. Internal derangement of TMJ (ant. Disc displacement with reduction)
4. Localized TMJ pain

Criteria of exclusion:

1. Psychiatric illness
2. Previous TMJ surgery
3. Suffering from joint trauma
4. Cellulitis or severe laceration of pre-auricular skin covering TMJ

Intervention:

The patients divided into two groups. Group one contains 20 patients will be treated by arthrocentesis with lactate ringer only (control group). Group 2 contains 20 patients will be treated by arthrocentesis with lactate ringer followed by injection with piroxicam 2 ml (40mg) (study group). The patient should have done MRI shows internal derangement. Maximum mouth opening should be measured before procedure.

Arthrocentesis technique will be done under aseptic condition using betadine (betadine: /7.5/m/v povidone iodine USP Nile Company, under license by Switzerland), auriculotemporal nerve block anesthesia was included using carpule of mepivacaine (mepivacaine HCL2% with levonordefrin 1:20000, Alexandria Co. Pharmaceuticals, Alexandria, Egypt) and field infiltration at sites of joint penetration. External auditory canal is protected from accumulation of blood and fluid by a cotton pellet. A line should be drowned from outer canthus of the eye to ear tragus (canthal tragus line). The first needle (inlet) corresponding to glenoid fossa should be placed 1 cm from mid tragus and 2mm below canthal tragus line. The second needle (outlet) related to articular eminence should be placed 1cm from first needle and 1 cm below canthal tragus line. 20-gauge needle was introduced to posterior aspect of glenoid fossa first mark (inlet) and 18-gauge needle is introduced into second mark (outlet). 200ml of lactate ringer solution is introduced into inlet syringe the joint is manipulated by closing opening lateral movement and protrusion to allow flow of solution and release of adhesions and inflammatory mediators. Then the lactate ringer is collected in kidney dish through the outlet syringe. This technique should be done in both groups (1&2). In group 2 only after this procedure is done, we use the first needle in injection of 2 ml (40mg) piroxicam (feldene:1 ml ampoule piroxicam manufactured by Pfizer S.A.E) into the joint space. After injection is done the joint should be manipulated in different directions.

After the procedures for both groups postoperative medication should be prescribed which is antibiotics. Post-operative instruction should be followed. Which is soft diet and home physical therapy containing application of moist heat and mandibular exercise as opening, closing, protrusion, extrusion and lateral movement 4 times per day. 8 Data collection: data will be collected twice inter examiner relatability. Measurements and assessment: Follow-up for the first day there may be numbness around the auricle which affect hearing sensation end by the end of local anesthetic effect. Also, edema may occur which need prescription of antiedematous and anti inflammatory. then follow up after 1 week then after 2 weeks then after month then after 3 months then after 6 months. In the follow up we must notice the maximum mouth opening without pain, lateral excursion during opening and closing mouth and visual analogue scale of pain.

Statistics: independent simple T-test. Ethics: the study is approved by ethical committee of Ain Shams University and the patients sign informed consent after the procedures have been described in details.

ELIGIBILITY:
Inclusion Criteria:

1. Age range 18-60 years both gender 2. Patient have gone on noninvasive therapy (occlusal stent) for three months without good prognosis 3. Internal derangement of TMJ (ant. Disc displacement with reduction) 4. Localized TMJ pain

-

Exclusion Criteria:

* 1. Psychiatric illness 2. Previous TMJ surgery 3. Suffering from joint trauma 4. Cellulitis or severe laceration of pre-auricular skin covering TMJ

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — biological females
Enrollment: 40 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
mouth opening | six months
  un assited mouth opening in mm

CONTACTS AND LOCATIONS:
Locations (1):
- Ain shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
based on publication requirment

REFERENCES:
- [Result] Baruffi S, Saber AY, Martins T, Varacallo MA. Shoulder Arthrocentesis Technique. 2023 Aug 4. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK519052/ PMID 30085594